CLINICAL TRIAL: NCT05954481
Title: Evaluation of the Value of Measuring Pulmonary Arterial Pressures During Exercise in Hereditary Haemorrhagic Telangiectasia Patients With Hepatic Involvement - Pilot Study
Brief Title: Stress-Echography in Hereditary Haemorrhagic Telangiectasia Patient With Hepatic Involvement
Acronym: ROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL22_0487
Record Dates: First submitted 2023-07-13; First posted 2023-07-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Rendu Osler Disease
Keywords: HHT; Stress echography; Pulmonary arterial pressures
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HHT patients with hepatic involvement and high cardiac index (Other): HHT patients with a dilated (diameter > 6mm) or tortuous hepatic artery and an elevated cardiac index (> 3.5 l/mn/m²)
  Interventions: Other: Stress echocardiography
- HHT patients with hepatic involvement and normal cardiac index (Other): HHT patients with a dilated or tortuous hepatic artery and a normal cardiac index
  Interventions: Other: Stress echocardiography

INTERVENTIONS:
Other: Stress echocardiography — After a rest trans thoracic echocardiography (usual follow-up), eligible patients will have a stress ultrasound echocardiography on a dedicated cycle ergometer

SUMMARY:
The hepatic involvement of HHT (Hereditary Haemorrhagic Telangiectasia) disease is characterised by the formation of arterio-sus-hepatic shunts which lead to dilatation of the hepatic artery and may result in high output heart failure. This evolves silently for long-standing period from left ventricular cavities dilatation to advanced heart failure with post-capillary pulmonary hypertension (PH) (more rarely pre-capillary), and its evolution is poorly understood. The specific treatment options for HHT disease are either the use of anti-angiogenic therapy (bevacizumab) or liver transplantation. As rest echocardiography can only detect advanced cases or heart failure with rest PH, the investigators speculate that exercise echocardiography can provide additional information in patients without rest PH. The hypothesis is that an exaggerated pulmonary pressure increase during exercise may precede the occurrence of rest PH in the course of the disease. It could identify patients with substantial heart failure at an earlier stage and may facilitate the access to liver transplantation. These parameters have never been studied in this context and it seems interesting to evaluate them in this pilot study.

The investigators hypothesise that HHT (Hereditary Haemorrhagic Telangiectasia) patients with hepatic involvement and cardiac high output will have significantly greater and/or earlier elevation of exercise pulmonary arterial pressures than those with normal cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* HHT patient > 18 yo
* Hepatic involvement (hepatic artery diameter > 6mm)
* Patient having received the information and signed the informed consent form
* Patient affiliated to a social security scheme or beneficiaries of a similar scheme

Exclusion Criteria:

* Haemoglobin < 90 g/L
* Active Infection
* Atrial Fibrillation permanent or persistent
* Known cardiopathy
* Pregnant or breastfeeding woman (by questioning)
* Adult subject to a legal protection measure (guardianship)
* Participation in another clinical trial that may interfere with the proposed trial (investigator judgment)
* Patient physically unable to pedal
* Patient with Pulmonary arteriovenous malformations awaiting embolization
* Patient treated with beta-blockers

Secondary Exclusion Criteria verified on rest ultrasound

* PAH (Pulmonary Arterial Hypertension) at rest (Vmax > 2.8 m/sec)
* Inability to obtain a stream of IT at rest
* Patient with atrial fibrillation (AF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Comparison of exercise pulmonary artery systolic pressure in patients with HHT and liver involvement. | Day 1
  The systolic pulmonary artery pressure (PAPS) during exercise will be compared between the two groups of patients. PAPS will be estimated by the maximum velocity (Vmax) of tricuspid insufficiency flow at peak exercise on cardiac ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille BERGEROT, MD, Principal Investigator — Service d'Explorations fonctionnelles cardiovasculaires - Hôpital Louis Pradel - HCL
Locations (2):
- France (2):
  - Service Explorations fonctionnelles cardiovasculaires - Hôpital Louis Pradel, Bron
  - Service génétique - Hôpital Femme Mère Enfant, Bron

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dr. Cyrille Bergerot Co-Authors: Sophie Dupuis-Girod, MD; Alexandre Guilhem, MD; Thomas Barret, MD; Quentin Barrier, MD; Anne Emmanuelle Fargeton; Helene Thibault, MD, PhD. Exercise Pulmonary Arterial Pressure during Exercise Stress Echocardiography in Hereditary Hemorrhagic Telangiectasia. International Journal of Cardiology.